CLINICAL TRIAL: NCT04404686
Title: Vaginal Indomethacin Versus Oral Nifedipine for Preterm Labor; a Randomized Controlled Trial
Brief Title: Vaginal Indomethacin for Preterm Labor
Acronym: TOCOMED
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Sheba Medical Center (Other Government); Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Hila Hocler MD, Principal Investigator, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOCOMED-HMO-CTIL
Record Dates: First submitted 2020-05-07; First posted 2020-05-27 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Obstetric Labor, Premature
Keywords: preterm labor; tocolysis; prematurity
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Indomethacin; Nifedipine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Caregivers will receive a closed envelope with the drug to be used. since the routes of administration are different, from that point on the caregiver and patient will be aware of chosen drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Indomethacin group (Experimental): Group of patients receiving Indomethacin for preterm labor treatment.
  Interventions: Drug: Indomethacin
- Nifedipine group (Active Comparator): Group of patients receiving Nifedipine for preterm labor treatment.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Indomethacin — Per vagina administration of 100 mg followed by a second 100 mg dosage the following day
  Other Names: Indomed
  Arms: Indomethacin group
Drug: Nifedipine — Per os administration according to current protocol of 20mg each 20 minutes for 1 hour followed by 20 mg q8 for 48 hours.
  Other Names: Pressolat
  Arms: Nifedipine group

SUMMARY:
Indometacin is a cyclooxygenase agent from the NSAID family that has been used to treat preterm contractions since the 70's by preventing the synthesis of prostaglandins. It has been shown to be significantly more effective than placebo and postpone labor for 7-10 days, prolong pregnancies above 37 weeks of gestation and reduce numbers of small for gestational age neonates.

Nifedipine is a calcium channel blocker agent that has been shown to reduce rates of labor within 48 hours from treatment.

Previous studies comparing rectal Indometacin to oral nifedipine were inconclusive.

Prostaglandins are synthesized in the uterus and the uterine cervix and therefore local administration of Indometacin may be more effective than other forms of administration, as been shown in a previous study.

In this study we aim to compare vaginal Indometacin administration to a commonly used tocolytic agent, nifedipine.

ELIGIBILITY:
Inclusion Criteria:

* Singe fetus
* Gestational age between 24+0/7 and 31+6/7
* At least one uterine contraction in ten minutes for at least 20 minutes upon tocography admission
* Cervical parameters: 1 cm dilation or more or 80% cervical effacement or cervical length 20mm or less

Exclusion Criteria:

* Rupture of membranes
* Vaginal bleeding
* Cervical dilation ≥5cm
* Known fetal malformations
* Fetal heart rate abnormalities
* Suspected placental abruption of adherent placental syndrome
* Known sensitivity to one of the drugs used in the study (Indometacin and nifedipine)
* Maternal hypotension and known aortic or mitral stenosis
* Presence of cervical cerclage
* Previous administration of tocolytic drugs in current pregnancy

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Enrollment: 300 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Time to delivery | through study completion, approximately 1 year
  The time from administration of intervention do delivery
Gestational age | through study completion, approximately 1 year
  Days from last menstrual period

SECONDARY OUTCOMES:
Rate of preterm deliveries | through study completion, approximately 1 year
  Rate of deliveries under 37+0/7 weeks of gestation
Rate of remote from term deliveries | through study completion, approximately 1 year
  Rate of deliveries under 34+0/7 weeks of gestation
Rate of extreme preterm deliveries | through study completion, approximately 1 year
  Rate of deliveries under 28+0/7 weeks of gestation
neonatal immediate outcomes | through study completion, approximately 1 year
  Neonatal Apgar scores
Neonatal immediate outcome | through study completion, approximately 1 year
  Neonatal umbilical cord pH levels
Neonatal birth weight | through study completion, approximately 1 year
  birth wight as recorded in chart in grams
Neonatal outcomes | through study completion, approximately 1 year
  neonatal intensive care unit administration rate

CONTACTS AND LOCATIONS:
Overall Officials: Hila Hochler, MD, Principal Investigator — Hadassah Medical Organization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niebyl JR, Blake DA, White RD, Kumor KM, Dubin NH, Robinson JC, Egner PG. The inhibition of premature labor with indomethacin. Am J Obstet Gynecol. 1980 Apr 15;136(8):1014-9. doi: 10.1016/0002-9378(80)90629-8. PMID 7369252
- [Background] Zuckerman H, Shalev E, Gilad G, Katzuni E. Further study of the inhibition of premature labor by indomethacin. Part II double-blind study. J Perinat Med. 1984;12(1):25-9. doi: 10.1515/jpme.1984.12.1.25. PMID 6374098
- [Background] Besinger RE, Niebyl JR, Keyes WG, Johnson TR. Randomized comparative trial of indomethacin and ritodrine for the long-term treatment of preterm labor. Am J Obstet Gynecol. 1991 Apr;164(4):981-6; discussion 986-8. doi: 10.1016/0002-9378(91)90569-d. PMID 2014850
- [Background] Haas DM, Imperiale TF, Kirkpatrick PR, Klein RW, Zollinger TW, Golichowski AM. Tocolytic therapy: a meta-analysis and decision analysis. Obstet Gynecol. 2009 Mar;113(3):585-594. doi: 10.1097/AOG.0b013e318199924a. PMID 19300321
- [Background] O'Brien WF. The role of prostaglandins in labor and delivery. Clin Perinatol. 1995 Dec;22(4):973-84. PMID 8665768
- [Background] Bry K, Hallman M. Prostaglandins, inflammation, and preterm labor. J Perinatol. 1989 Mar;9(1):60-5. PMID 2496208
- [Background] Abramov Y, Nadjari M, Weinstein D, Ben-Shachar I, Plotkin V, Ezra Y. Indomethacin for preterm labor: a randomized comparison of vaginal and rectal-oral routes. Obstet Gynecol. 2000 Apr;95(4):482-6. doi: 10.1016/s0029-7844(99)00578-5. PMID 10725476
- [Background] Flenady V, Wojcieszek AM, Papatsonis DN, Stock OM, Murray L, Jardine LA, Carbonne B. Calcium channel blockers for inhibiting preterm labour and birth. Cochrane Database Syst Rev. 2014 Jun 5;2014(6):CD002255. doi: 10.1002/14651858.CD002255.pub2. PMID 24901312
- [Background] Reinebrant HE, Pileggi-Castro C, Romero CL, Dos Santos RA, Kumar S, Souza JP, Flenady V. Cyclo-oxygenase (COX) inhibitors for treating preterm labour. Cochrane Database Syst Rev. 2015 Jun 5;2015(6):CD001992. doi: 10.1002/14651858.CD001992.pub3. PMID 26042617
- [Background] Kashanian M, Bahasadri S, Zolali B. Comparison of the efficacy and adverse effects of nifedipine and indomethacin for the treatment of preterm labor. Int J Gynaecol Obstet. 2011 Jun;113(3):192-5. doi: 10.1016/j.ijgo.2010.12.019. Epub 2011 Apr 1. PMID 21457979
- [Background] Klauser CK, Briery CM, Keiser SD, Martin RW, Kosek MA, Morrison JC. Effect of antenatal tocolysis on neonatal outcomes. J Matern Fetal Neonatal Med. 2012 Dec;25(12):2778-81. doi: 10.3109/14767058.2012.714819. Epub 2012 Aug 20. PMID 22873356
- [Background] Klauser CK, Briery CM, Martin RW, Langston L, Magann EF, Morrison JC. A comparison of three tocolytics for preterm labor: a randomized clinical trial. J Matern Fetal Neonatal Med. 2014 May;27(8):801-6. doi: 10.3109/14767058.2013.847416. Epub 2013 Oct 11. PMID 24090282
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046